CLINICAL TRIAL: NCT03851835
Title: Multi-dose Oral Ondansetron For Pediatric Gastroenteritis: A Pragmatic Randomized Controlled Trial
Brief Title: Multi-DOSE Oral Ondansetron for Pediatric Acute GastroEnteritis
Acronym: DOSE-AGE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Women and Children's Health Research Institute (WCHRI) (Unknown); The Hospital for Sick Children (Other); Children's Hospital Research Institute of Manitoba (Other); University of Manitoba (Other); Université de Montréal (Other); University of Ottawa (Other); University of Alberta (Other); Alberta Children's Hospital Research Institute (Other); Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OND18-2045
Record Dates: First submitted 2019-02-19; First posted 2019-02-22 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Acute Gastroenteritis; Viral Illness; Vomiting; Diarrhea
Keywords: Vomiting; Zofran; Ondansetron; Gastroenteritis; Pediatrics; DOSE-AGE
MeSH Terms: conditions — Virus Diseases; Vomiting; Diarrhea; Gastroenteritis | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ondansetron Oral Solution (Experimental): Ondansetron Oral Solution (4mg/5mL solution) - Dose = 0.15mg/kg. One dose every 8 hours (q8h), as needed. Up to a maximum of six doses over 48 hours.
  Interventions: Drug: Ondansetron Oral Solution
- Placebo Oral Solution (Placebo Comparator): Compounded Placebo Oral Solution to match experimental arm
  Interventions: Drug: Oral Placebo

INTERVENTIONS:
Drug: Ondansetron Oral Solution — Six doses of oral ondansetron (0.15mg/kg) to be administered q8h (every 8 hours) to a maximum of 3 times in a 24 hour period, are provided to the participant/caregiver for use after emergency department disposition (i.e. home use), as needed.
  Other Names: Zofran
  Arms: Ondansetron Oral Solution
Drug: Oral Placebo — Six doses of oral placebo (0.15mg/kg) to be administered q8h (every 8 hours) to a maximum of 3 times in a 24-hour period, are provided to the participant/caregiver for use after emergency department disposition (i.e. home use), as needed.
  Arms: Placebo Oral Solution

SUMMARY:
A phase III, double-blind, parallel-design, randomized, placebo-controlled trial to compare multi-dose oral Ondansetron with placebo as treatment for vomiting secondary to acute gastroenteritis (AGE), after Emergency Department discharge.

DETAILED DESCRIPTION:
The annual burden of acute gastroenteritis in the United States includes 17 million related episodes and 473,832 hospitalizations. Although oral-rehydration therapy is recommended for children with mild-to-moderate dehydration, it has historically been underused with emergency department (ED) clinicians being more likely to choose intravenous over oral rehydration especially when vomiting is a major symptom. In fact, nearly 95% of children undergoing oral rehydration in Canadian EDs present with recent vomiting. To address this issue, the investigators conducted both a landmark clinical trial and a recent meta-analysis that have demonstrated that the ED use of ondansetron, an anti-emetic, leads to reductions in intravenous rehydration and hospitalization and is cost-effective. However, the available data revealed some associations with increased diarrhea and no evidence of benefits associated with ongoing ondansetron use following ED discharge. Despite the lack of available data, the provision of multiple doses of ondansetron for home use has become routine in many EDs across North America. The literature has differing opinions on the topic of ongoing ondansetron use after ED discharge and given the limited evidence supporting its use, the potential side effects and additional cost, there is an urgent need to definitively evaluate the effect of multiple doses of ondansetron in children, focusing on family-centred, post-index visit outcomes.

A phase III, double-blind, parallel-design, randomized, placebo controlled trial to compare multi-dose oral Ondansetron with placebo as treatment for vomiting secondary to acute gastroenteritis (AGE), after Emergency Department discharge will be conducted. Children and youth, age 6 months to 17.99 years will be enrolled at six (6) Canadian Emergency Departments. The total number of participants recruited will be 1030. Participants will be enrolled at six (6) pediatric emergency departments across Canada.

Children who are provided a minimum of one dose of ondansetron as part of their routine clinical care AND meet other eligibility criteria will be randomized to receive an at-home kit with six (6) doses of Ondansetron Hydrochloride Dihydrate Oral Solution (4mg/5mL solution; dosed at 0.15mg/kg to a maximum single dose of 8mg) or equivalent volume in a Placebo Oral Solution to be administered no sooner than 8 hours after the initial clinical dose was provided by the ED physician. Over the subsequent 48 hours, the study intervention will be administered at a rate of 1 dose every 8 hours (q8h) to a maximum of 3 doses a day (in a 24-hour period (TID)) at the caregiver's discretion. Two (2) additional doses will be provided to the caregiver in case the child vomits a dose.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to comply with all study procedures and availability for the duration of the study.
* Diagnosis of acute intestinal infectious process (as defined by the protocol) confirmed. by the treating physician.
* Age 6 months to 17.99 years.
* Presence of ≥ 3 episodes of vomiting in the preceding 24-hour period.
* Duration of vomiting and/or diarrheal symptoms < 72 hours.
* A minimum of 1 episode of vomiting within 6 hours of the screening process performed by the research team.
* A minimum of 1 dose of ondansetron (oral or intravenous) provided during the current emergency department visit.

Exclusion Criteria:

* Bilious or bloody vomit during current illness.
* Known hypersensitivity to ondansetron or any serotonin receptor antagonist (e.g. palonosetron, dolasetron, granisetron).
* Known allergic reaction to components of ondansetron (citric acid, sodium benzoate, sodium citrate dihydrate, and strawberry flavor, sorbitol) or the placebo medication (methylparaben, glycerin, citric acid, potassium sorbate, sorbitol, strawberry flavor).
* History or family history (first degree relative) of prolonged QT syndrome.
* Presence of complex congenital heart disease.
* History or family history (first degree relative) of cardiac arrhythmia.
* Concomitant use (within the past 48 hours) of any of the following: QTc prolonging medications, medications known to cause torsades de pointes, medications that cause electrolyte abnormalities, serotonergic or neuroleptic medications, or any 5-HT3 receptor antagonist excluding ondansetron.
* Unable to complete follow-up.
* Previously enrolled in this study.
* History or family history of G6PD deficiency.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1030 (Actual)
Dates: Start 2019-09-14 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2024-07-06 (Actual)

PRIMARY OUTCOMES:
Development of moderate to severe disease as defined by the Modified Vesikari Scale (MVS) Score of ≥ 9 following ED evaluation - change in the MVS score between Hour 0 and Hour 168 of the study. | Measured 24, 48, and 168 hours after baseline visit
  The Modified Vesikari Scale Score (MVS) is a composite measure which includes several variables representing the severity of disease - points are summed to provide an overall score:
  * Duration of diarrhea (hours): 0 (0 points), 1-96 (1 point), 97-120 (2 points), ≥121 (3 points)
  * Maximum number of watery stools per 24 hour period: 0 (0 points), 1-3 (1 point), 4-5 (2 points), ≥6 (3 points)
  * Duration of vomiting (hours): 0 (0 points), 1-24 (1 point), 25-48 (2 points), ≥49 (3 points)
  * Maximum number of vomiting episodes per 24 hour period: none (0 points), 1 (1 point), 2-3 (2 points), ≥5 (3 points).
  * Maximum recorded rectal temperature (degrees Celsius): <37.0 (0 points), 37.1-38.4 (1 point), 38.5-38.9 (2 points), ≥39.0 (3 points)
  * Unscheduled health care visit: None (0 points), Primary Care (2 points), emergency department (3 points)
  * Treatment: None (0 points), Rehydration with IV fluids (1 point), Hospitalization (2 points)

SECONDARY OUTCOMES:
Vomiting Duration | Measured 24, 48, and 168 hours after baseline visit
  Number of hours of vomiting following ED disposition.
Vomiting Frequency | Measured 24, 48, and 168 hours after baseline visit
  Number of episodes of vomiting following ED disposition.
Vomiting Proportion | Measured 24, 48, and 168 hours after baseline visit
  The proportion who experience vomiting following ED disposition.
Proportion of participants who require an unscheduled health care visit | Measured 24, 48, and 168 hours after baseline visit
  Unscheduled health care provider visits following Emergency Department disposition. Is there a difference in the proportion who require an unscheduled health care provider visit following ED disposition.
Proportion of participants who require Intravenous (IV) Rehydration | Measured 24, 48, and 168 hours after baseline visit
  Is there a difference in the proportion who require intravenous rehydration following ED disposition.
Satisfaction with care: 5 point Likert Scale | 168 hours after baseline
  Caregivers will be asked about their level of satisfaction with the therapy provided measured on the following 5 point Likert scale (choose one option):
  * 1 - Very dissatisfied
  * 2 - Dissatisfied
  * 3 - Neither satisfied, nor dissatisfied
  * 4 - Satisfied
  * 5 - Very Satisfied

OTHER OUTCOMES:
Safety Profile of Multiple Doses of Oral Ondansetron | Measured 24, 48, and 168 hours after baseline visit
  To determine if the discharge of children with AGE associated vomiting who are administered ondansetron in the ED with additional doses to be taken at home is associated with adverse events (e.g. diarrhea, revisits) as compared with placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Freedman, MD, Principal Investigator — University of Calgary
Locations (6):
- Canada (6):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - Children's Hospital of Winnipeg, Winnipeg, Manitoba
  - Children's Hospital London Health Sciences Centre, London, Ontario
  - Children's Hospital of Eastern Ontario (CHEO), Ottawa, Ontario
  - Centre Hospitalier Universitaire Sainte Justine, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Freedman SB, Williamson-Urquhart S, Plint AC, Dixon A, Beer D, Joubert G, Pechlivanoglou P, Finkelstein Y, Heath A, Zhang JZ, Wallace A, Offringa M, Klassen TP; Pediatric Emergency Research Canada Innovative Clinical Trials Study Group. Multidose Ondansetron after Emergency Visits in Children with Gastroenteritis. N Engl J Med. 2025 Jul 17;393(3):255-266. doi: 10.1056/NEJMoa2503596. PMID 40673584
- [Derived] Heath A, Rios JD, Williamson-Urquhart S, Pechlivanoglou P, Offringa M, McCabe C, Hopkin G, Plint AC, Dixon A, Beer D, Gouin S, Joubert G, Klassen TP, Freedman SB; PERC-KIDSCAN DOSE-AGE Study Group. A pragmatic randomized controlled trial of multi-dose oral ondansetron for pediatric gastroenteritis (the DOSE-AGE study): statistical analysis plan. Trials. 2020 Aug 24;21(1):735. doi: 10.1186/s13063-020-04651-1. PMID 32838813
- [Derived] Freedman SB, Williamson-Urquhart S, Heath A, Pechlivanoglou P, Hopkin G, Gouin S, Plint AC, Dixon A, Beer D, Joubert G, McCabe C, Finkelstein Y, Klassen TP; KidsCAN-Pediatric Emergency Research Canada (PERC) Innovative Pediatric Clinical Trials DOSE-AGE Study Group. Multi-dose Oral Ondansetron for Pediatric Gastroenteritis: study Protocol for the multi-DOSE oral ondansetron for pediatric Acute GastroEnteritis (DOSE-AGE) pragmatic randomized controlled trial. Trials. 2020 May 27;21(1):435. doi: 10.1186/s13063-020-04347-6. PMID 32460879